CLINICAL TRIAL: NCT03982498
Title: Diagnostic Accuracy of Increased Serum Cytokine Levels as a Marker of Paralytic Ileus Following Robotic Radical Cystectomy
Brief Title: Cytokine-guided Robotic Cystectomy
Acronym: CY-ROC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: University of Hertfordshire (Other)
Responsible Party: Sponsor
Other Study IDs: RD2018-65
Record Dates: First submitted 2019-06-09; First posted 2019-06-11 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a recognised complication of surgery known as a 'Paralytic Ileus', where bowel function is reduced after an operation, causing an obstruction and resulting in nausea and vomiting. This complication is more common in patients that have robotic surgery due to the positioning required and the gas pressures required for keyhole/robotic surgery. While some of the factors involved in a paralytic ileus are known, the full mechanism and the chemicals involved are not yet fully understood.

This study is looking at the level of specific chemicals called 'cytokines', and the changes in the level of these cytokines in the blood before and after robotic surgery, specifically during bladder removal (cystectomy). Cytokine levels will be compared against post-operative recovery and whether a paralytic ileus is developed.

DETAILED DESCRIPTION:
Cytokines are signalling proteins that are release by immune cells in response to stress on the body. In this study the aim is to evaluate the concordance between cytokine rise (specifically monitoring the following cytokines: Interferon (IFN)-gamma, tumour necrosis factor (TNF)-alpha, Interleukin (IL) -1beta, IL-2, IL-4, IL-6, IL-12 and IL-17) and postoperative ileus (a condition where bowel function slows causing build up of faecal matter) following robotic radical cystectomy and the pneumoperitoneum (gas insufflation of the abdomen) pressures that were required intra-operatively.

This study includes patients undergoing radical cystectomy. The study will measure pre-anaesthetic, post-anaesthetic, immediately post-operatively and two further post-operative serum cytokines levels and compare them with the pneumoperitoneal pressures required intra-operatively and the outcome of whether a clinical diagnosis of paralytic ileus was made.

Serum cytokine levels will be taken on five occasions:

1. st Sample (Baseline)-Before induction of anaesthetic
2. nd Sample-Immediately after induction of anaesthetic
3. rd Sample-Immediately post-operative
4. th Sample - 2 hours post-operative
5. th Sample - 1 day post-operative

No alterations will be made to the care of the patient, this is purely an observational study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 40 and 75 years of age
* Patients undergoing a Robotic radical cystectomy
* Patient consenting to enter the study
* Patients consenting for blood samples for cytokine analysis

Exclusion Criteria:

* Patients <40 years of age and patients >75 years of age
* Patients unwilling or unable to consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing planned robotic radical cystectomy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-06-14 (Estimated); Study Completion 2022-06-14 (Estimated)

PRIMARY OUTCOMES:
Correlation between cytokine rise (intra-and post-operatively) and postoperative ileus following robotic radical cystectomy | 24 hours post-surgery
  Serum cytokine levels

CONTACTS AND LOCATIONS:
Locations (1):
- East and North Hertfordshire NHS Trust, Stevenage, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No